CLINICAL TRIAL: NCT00888537
Title: Wiser Choices in Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nilay D. Shah, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-000748
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Decision aid; Heart attack; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Experimental): Patients in this arm will discuss medications to help the heart heal after a heart attack with the clinician and the help of the acute myocardial infarction (AMI) Choice Decision Aid.
  Interventions: Other: AMI Choice Decision Aid
- Usual Care (Active Comparator): Patients and clinicians in this arm will discuss medications to help the heart heal after a heart attack in their usual manner.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: AMI Choice Decision Aid — The decision aid describes the risk of dying in the first six months following a heart attack without and with taking a bundle of medications to help the heart heal.
  Arms: Decision Aid
Other: Usual Care — Patients and clinicians in this arm will discuss medications to help the heart heal after a heart attack in their usual manner.
  Arms: Usual Care

SUMMARY:
Patients who are hospitalized because of a heart attack are prescribed a number of medicines to help the heart heal. The investigators will examine different ways in which clinicians share information about those treatment options with patients and the impact that this can have on patients' choices and health.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 90
* Hospitalized at Saint Marys Hospital
* A primary diagnosis of AMI,
* Have heart rate, blood pressure, troponin and creatinine measurements,
* There is an intention to offer treatment medications
* Are able and willing to provide informed consent

Exclusion Criteria:

* Have not had a myocardial infarction
* Have significant cognitive, visual impairment,
* Non-English speaker
* Have a Do Not Intubate/Do Not Resuscitate (DNI/DNR) status
* Will be discharged to a nursing home
* AMI is not the presumptive diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Increases adherence to cardiac medications with proven benefits | 6 months
Reduces patients' decisional conflict (increase patient decisional quality) | During hospital stay
Decreases rehospitalization rates and death | 5 weeks and 6 months
Increase patient knowledge of medication to help the heart heal | During hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ting, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Saint Marys Hospital, Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Branda ME, Kunneman M, Meza-Contreras AI, Shah ND, Hess EP, LeBlanc A, Linderbaum JA, Nelson DM, Mc Donah MR, Sanvick C, Van Houten HK, Coylewright M, Dick SR, Ting HH, Montori VM. Shared Decision-Making for Patients Hospitalized with Acute Myocardial Infarction: A Randomized Trial. Patient Prefer Adherence. 2022 Jun 1;16:1395-1404. doi: 10.2147/PPA.S363528. eCollection 2022. PMID 35673524
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289